CLINICAL TRIAL: NCT01534208
Title: An Open Label, Escalating Dose, 6 Month Phase III Safety Study Of Enclomiphene Citrate in the Treatment of Men With Secondary Hypogonadism
Brief Title: Safety Study of Enclomiphene Citrate in the Treatment of Men With Secondary Hypogonadism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZA-300
Record Dates: First submitted 2012-02-09; First posted 2012-02-16 (Estimated); Results first posted 2014-07-24 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-06

CONDITIONS: Secondary Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Enclomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Androxal 12.5 mg (Experimental): Androxal 12.5 mg daily
  Interventions: Drug: Androxal
- Androxal 25 mg (Experimental): Androxal 25 mg daily
  Interventions: Drug: Androxal

INTERVENTIONS:
Drug: Androxal — Androxal, oral, 12.5 mg capsule, taken once daily. Dose may be increased from 12.5 mg to 25 mg if indicated
  Other Names: Enclomiphene citrate

SUMMARY:
ZA-300 is meant to determine the safety profile of Androxal (enclomiphene citrate) in men with secondary hypogonadism.

DETAILED DESCRIPTION:
This study is a phase III, open label safety study with a six month active dosing period. All subjects will be started at 12.5 mg Androxal and titrated to 25 mg if needed. Safety will be assessed by physical and visual acuity exams, slit lamp eye exams, clinical laboratory tests and adverse event reporting.

ELIGIBILITY:
Inclusion Criteria:

1. Secondary hypogonadal males between the ages of 18 and 65
2. Men currently using topical testosterone products should wash-out for at least 7 days before Visit 1.
3. All clinical laboratory tests within normal ranges (any clinically significant deviation of laboratory results will require approval of sponsor)
4. Previously or concurrently diagnosed as having secondary hypogonadism and confirmed with morning testosterone level < 350 ng/dL for men age < 55 and < 300ng/dl for men age 55-65
5. LH < 15mIU/mL (at Visit 1 only)
6. Ability to complete the study in compliance with the protocol
7. Ability to understand and provide written informed consent.

Exclusion Criteria:

1. Use of an injectable pelleted testosterone within 6 months prior to study (men currently on topical testosterone products may be enrolled in the study after a 7-day washout period).
2. Use testosterone injection, spironolactone, cimetidine, Clomid, 5α-reductase inhibitors, hCG, androgen, estrogen, anabolic steroid, DHEA, or herbal hormone products during the study
3. Use of Clomid in the past year
4. Uncontrolled hypertension based on the Investigator's assessment at baseline. Subjects treated for Type II diabetes will be allowed into the study.
5. A hematocrit ≥ 51% or a hemoglobin ≥ 17 g/dL
6. Clinically significant abnormal findings on screening examination, based on the Investigator's assessment.
7. Use of an investigational drug or product, or participation in a drug or medical device research study within 30 days prior to receiving study medication.
8. Known hypersensitivity to Clomid
9. Symptomatic cataracts (nuclear sclerosis cataract or cortical cataract grade > 2 based on 0-4 scale or any trace of posterior subcapsular cataract)
10. Any condition which in the opinion of the investigator would interfere with the participant's ability to provide informed consent, comply with study instructions, possibly confound interpretation of study results, or endanger the participant if he took part in the study
11. Irreversibly infertile or compromised fertility (cryptorchism, Kallman Syndrome, primary hypogonadism, or tumors of the pituitary)
12. Current or history of breast cancer
13. Current or history of prostate cancer or a suspicion of prostate disease unless ruled out by prostate biopsy, or a PSA > 3.6
14. Presence or history of known hyperprolactinemia with or without a tumor
15. Chronic use of medications use such as glucocorticoids
16. Chronic use of narcotics
17. Subjects know to be positive for HIV
18. End stage renal disease
19. Subjects with cystic fibrosis (mutation of the CFTR gene)
20. Enrollment in a previous Androxal study

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 499 (Actual)
Dates: Start 2012-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph S Podolski, Study Chair — Repros Therapeutics Inc.
Locations (29):
- United States (29):
  - Clinical Research Advantage, Glendale, Arizona
  - Clinical Research Advantage, Phoenix, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Catalina Research Institute, Chino, California
  - SC Clinical Research, Garden Grove, California
  - South Orange County Endocrinology, Laguna Hills, California
  - Anthony Mills, MD, Los Angeles, California
  - SD Uro-Research, San Diego, California
  - San Diego Sexual Medicine, San Diego, California
  - SC Clinical Research, Santa Ana, California
  - West Coast Clinical Research, Tarzana, California
  - Clinical Research Advantage, Colorado Springs, Colorado
  - Meridien Research, Bradenton, Florida
  - Florida Fertility Institute, Clearwater, Florida
  - Therafirst Medical Center, Fort Lauderdale, Florida
  - East Coast Institute for Clinical Research, Jacksonville, Florida
  - East Coast Institute for Research, Jacksonville, Florida
  - Well Pharma Medical Research, Miami, Florida
  - Cetero Research, Miami Gardens, Florida
  - DMI Research, Pinellas Park, Florida
  - Ebon Bourne, MD, Plantation, Florida
  - Meridien Research, St. Petersburg, Florida
  - IRC Clinics, Towson, Maryland
  - Premier Urology Associates, Lawrenceville, New Jersey
  - Advances in Health, Houston, Texas
  - Breco Research, Sugar Land, Texas
  - Center of Reproductive Medicine, Webster, Texas
  - Lone Peak Family Medicine, Draper, Utah
  - Granger Medical Clin ic, Riverton, Utah

REFERENCES:
- See also: Sponsor home page — http://www.reprosrx.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Androxal 12.5 mg: Androxal 12.5 mg daily
  Androxal, oral, 12.5 mg capsule, taken once daily
- Androxal 25 mg: Androxal 25 mg daily
  Androxal, oral, 25 mg capsule, taken once daily
Period: Overall Study
Arm/Group | Androxal 12.5 mg | Androxal 25 mg
Started | 216 | 283
Completed | 159 | 234
Not Completed | 57 | 49
Not completed — Lost to Follow-up | 19 | 14
Not completed — Withdrawal by Subject | 6 | 20
Not completed — Adverse Event | 15 | 8
Not completed — Physician Decision | 2 | 0
Not completed — Lack of Efficacy | 0 | 3
Not completed — Protocol Violation | 2 | 2
Not completed — Sponsor decision | 4 | 1
Not completed — Subject relocation | 2 | 0
Not completed — Lab assessment | 2 | 1
Not completed — Eligibility error | 3 | 0
Not completed — PCP decision | 1 | 0
Not completed — Needed prohibited meds | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | Androxal 12.5 mg | Androxal 25 mg | Total
Number analyzed (Participants) | 216 | 283 | 499
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (8.5) | 49.5 (7.7) | 48.6 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 216 | 283 | 499
Region of Enrollment [Number; unit: participants]
  United States | 216 | 283 | 499

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Morning Testosterone at 26 Weeks
Description: Changes in values from baseline of total morning testosterone levels at Week 26
Time Frame: 6 months
Population: Intent to Treat population
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Androxal 12.5 mg | Androxal 25 mg
Number analyzed (Participants) | 168 | 242
ng/dL | 280.9 (141.4) | 214.7 (154.7)

2. Primary Outcome: Change From Baseline in LH
Description: Mean change from baseline in LH at end of treatment (26 weeks)
Time Frame: 6 months
Population: ITT
Measure: Mean (Standard Deviation); unit: mIu/mL
Arm/Group | Androxal 12.5 mg | Androxal 25 mg
Number analyzed (Participants) | 168 | 242
mIu/mL | 4.81 (5.69) | 4.27 (4.29)

3. Primary Outcome: Absolute Values of Morning Testosterone
Description: Absolute values of morning testosterone at end of treatment (26 weeks)
Time Frame: 6 months
Population: ITT
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Androxal 12.5 mg | Androxal 25 mg
Number analyzed (Participants) | 216 | 283
ng/dL | 511.6 (140.8) | 416.7 (154.7)

4. Primary Outcome: Mean Change From Baseline FPG
Description: Mean changes in Fasting Plasma Glucose from baseline to end of treatment (26 weeks)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Androxal 12.5 mg | Androxal 25 mg
Number analyzed (Participants) | 168 | 242
mg/dL | -5.4 (30.8) | -5.0 (29.3)

5. Primary Outcome: Change From Baseline in BMI
Description: Mean change from baseline in BMI at end of treatment (26 weeks)
Time Frame: 6 months
Population: ITT
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Androxal 12.5 mg | Androxal 25 mg
Number analyzed (Participants) | 216 | 283
kg/m2 | 0.2 (1.4) | 0.3 (1.1)

6. Primary Outcome: Change From Baseline in FSH
Description: Change from baseline in FSH at end of treatment (26 weeks)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Androxal 12.5 mg | Androxal 25 mg
Number analyzed (Participants) | 168 | 242
U/L | 5.20 (5.19) | 5.42 (5.48)

ADVERSE EVENTS:
Time Frame: From first administration of study drug until 8 weeks after end of treatment (8 months total)
Arm/Group | Androxal 12.5 mg | Androxal 25 mg
Serious Adverse Events (participants affected / at risk) | 6/207 | 9/283
Other Adverse Events (participants affected / at risk) | 66/207 | 92/283
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Androxal 12.5 mg (N=207) | Androxal 25 mg (N=283)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (2)
Food poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Kidney infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Seminoma (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Knee arthroplasy (Surgical and medical procedures) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Androxal 12.5 mg (N=207) | Androxal 25 mg (N=283)
Upper respiratory tract infection (Infections and infestations) | 26 (26) | 27 (27)
Headache (Nervous system disorders) | 12 | 23
Hot flush (General disorders) | 2 | 9
Influenza (Infections and infestations) | 7 | 5
Sinusitis (Infections and infestations) | 7 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 12
Dizziness (Nervous system disorders) | 6 | 5
Pollakiuria (Renal and urinary disorders) | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication, Investigator shall submit to the Sponsor a copy of any proposed publication. Sponsor shall have sixty (60) days to review the proposed publication for possible disclosure of Sponsor's Confidential Information and, upon request of Sponsor, Investigator shall delete any of Sponsor's Confidential Information or withhold submission of such publication to allow Sponsor to protect its intellectual property rights